CLINICAL TRIAL: NCT03783689
Title: The SNAP Trial: SPRINT® Peripheral Nerve Stimulation for the Treatment of Neuropathic Post-Amputation Pain in a Randomized, Double-blinded, Placebo-controlled, Multicenter Trial
Brief Title: The SNAP Trial: SPRINT® Peripheral Nerve Stimulation for the Treatment of Neuropathic Post-Amputation Pain
Acronym: SNAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic, Federal contract funding ended
Sponsor: SPR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0147-CSP-000
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Neuropathic Pain; Amputation
MeSH Terms: conditions — Neuralgia | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 (Treatment) (Active Comparator): Subjects in Group 1 will have Leads placed in the residual limb in the upper leg. These subjects will then use the SPRINT Peripheral Nerve Stimulation (PNS) System and will receive electrical stimulation for 8 weeks.
  Interventions: Device: SPRINT Peripheral Nerve Stimulation (PNS) System
- Group 2 (Control) (Sham Comparator): Subjects in Group 2 will have Leads placed in the residual limb in the upper leg. These subjects will then use the SPRINT Peripheral Nerve Stimulation (PNS) System and receive 8 weeks of sham stimulation. Subjects will then have the option to crossover and receive stimulation therapy.
  Interventions: Device: SPRINT Peripheral Nerve Stimulation (PNS) System

INTERVENTIONS:
Device: SPRINT Peripheral Nerve Stimulation (PNS) System — The SPRINT System delivers mild electrical stimulation to nerves in the residual limb. The SPRINT System includes two small wires (called "Leads") that are placed through the skin in the upper leg. It also includes a device worn on the body that delivers stimulation (called the SPRINT Stimulator).
  Other Names: SPRINT; SPRINT System

SUMMARY:
The purpose of this study is to determine if pain can be relieved by delivering small amounts of electricity (called "electrical stimulation") to the nerves in an individual's amputated leg.This study will involve the use of a Peripheral Nerve Stimulation (PNS) System that is made by SPR Therapeutics (the sponsor of the study). The PNS System was cleared by the FDA for up to 60 days of use for the management of chronic pain, including extremity (leg) pain.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 21 years old
* Lower extremity amputation
* Experiencing residual limb (stump) and/or phantom limb pain
* Healed amputation and healthy residual limb based upon the investigator's evaluation

Key Exclusion Criteria:

* Conditions with increased risk of infection (e.g., compromised immune system or history of recurrent skin infections)
* Implanted electronic device
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Pain Center of Arizona - Hope Research Institute, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - Lake Nona Medical Arts, Orlando, Florida
  - James A. Haley Veterans' Hospital, Tampa, Florida
  - Better Health Clinical Research, Newnan, Georgia
  - Northwestern University, Chicago, Illinois
  - Neuroscience Research Center, LLC, Overland Park, Kansas
  - OtriMed Clinical Research Center, Edgewood, Kentucky
  - MedVadis Research, Waltham, Massachusetts
  - Premier Pain Centers, Shrewsbury, New Jersey
  - Pain Management Center, Voorhees Township, New Jersey
  - Duke University, Durham, North Carolina
  - Center for Clinical Research, Winston-Salem, North Carolina
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After obtaining informed consent, subjects were evaluated for eligibility.
Groups:
- Group 1 (Treatment): Subjects in Group 1 were consented and met all eligibility criteria prior to randomization. These subjects had Leads placed in their residual limb and received electrical stimulation for up to 8 weeks via the SPRINT Peripheral Nerve Stimulation (PNS) System.
- Group 2 (Control): Subjects in Group 2 were consented and met all eligibility criteria prior to randomization. These subjects had Leads placed in their residual limb and received up to 8 weeks of sham stimulation. Three months after start of sham treatment, subjects were given the option to crossover and receive stimulation therapy via the SPRINT Peripheral Nerve Stimulation (PNS) System.
Period: Overall Study
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Started | 19 | 19
Safety Set (All subjects who were consented, randomized, and underwent Lead placement.) | 19 | 19
Full Analysis Set (Subjects who were consented, randomized, and continued to meet eligibility criteria prior to undergoing Lead placement.) | 18 | 18
Per Protocol Set (Subjects who were consented, randomized, continued to meet eligibility criteria prior to undergoing Lead placement, were implanted with at least one Lead, reported coverage of comfortable sensations in the target areas during weeks 5 to 8 post-start of treatment (SOT), have adequate diary completion for each qualifying region of pain, and continued eligibility during weeks 1 to 8 post-SOT.) | 13 | 16
Group 2 (Control Group Treatment Crossover) (Subjects who were consented, randomized to Group 2 (Control), received sham stimulation treatment, and crossed over to receive active stimulation treatment.) | 0 | 9
Completed | 10 | 14
Not Completed | 9 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Treatment) | Group 2 (Control) | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12.0) | 62.0 (10.5) | 59.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 15 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 17 | 18 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 14 | 15 | 29
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Employment Status [Count of Participants; unit: Participants]
  Currently Working | 3 | 4 | 7
  Retired (not due to health) | 4 | 4 | 8
  Unemployed | 1 | 1 | 2
  Student | 1 | 0 | 1
  Disabled / Retired (due to health) | 9 | 10 | 19
  Other (self-employed) | 1 | 0 | 1
Location of Amputation [Count of Participants; unit: Participants]
  Right Leg: Below Knee Amputation | 7 | 6 | 13
  Right Leg: Above Knee Amputation | 3 | 5 | 8
  Left Leg: Below Knee Amputation | 7 | 4 | 11
  Left Leg: Above Knee Amputation | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With ≥50% Reduction in Average Post-Amputation Pain (Residual Limb Pain [RLP] and/or Phantom Limb Pain [PLP])
Description: All subjects were asked to complete daily diaries to record their average residual limb pain and/or phantom pain intensities during the past 24 hours on each day of a 7-day period using an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average pain scores were calculated across the 7-day period for each region of pain at baseline and across weeks 5 to 8 post-start of treatment. Percent reduction was then calculated for each subject's qualifying region of pain (residual limb and/or phantom limb pain with qualifying average pain intensity at baseline). To be considered a success, subjects must have experienced ≥ 50% reduction in all qualifying regions of pain compared to their 7-day baseline diary average pain score(s). The number of successes is presented.
Time Frame: Baseline and 5 to 8 weeks post-start of treatment (SOT)
Population: Per Protocol Set presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 13 | 16
Participants | 6 | 3

2. Primary Outcome: Number of Subjects That Experienced at Least One Study-Related Adverse Event
Description: At each study visit following the baseline assessment at Visit 1, subjects were questioned if any changes in their medical status or condition have occurred since their previous visit. If the subject experienced a change that was a study-related adverse event, an Adverse Event Form was completed by the site. The number of subjects that experienced at least one study-related adverse event is reported here.
Time Frame: Up to 14 months for each Group 1 subject and up to 18 months for each Group 2 subject (time from baseline to last study visit)
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 19 | 19
Participants | 10 | 6

3. Secondary Outcome: Pain Interference
Description: Question 9 of the Brief Pain Inventory-Short Form (BPI-9) is a 7-part question that assesses the level of interference that subjects experience in their daily lives due to pain. The 7 categories are general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Subjects were asked to rate how much their post-amputation residual and/or phantom limb pains interfere with each aspect on an 11-point numerical scale where 0 represents "Does Not Interfere" and 10 represents "Completely Interferes." The average of these 7 scores was calculated for each subject at each time point. Percent reduction was then calculated for each subject's qualifying region of pain (residual limb and/or phantom limb pain with qualifying average pain intensity at baseline). To be considered a success, subjects must have experienced ≥ 50% reduction in all qualifying regions of pain compared to baseline. The number of successes is presented.
Time Frame: Visit 1 (Baseline), Visit 7 (4-weeks post-start of treatment [SOT]), Visit 11 (8-weeks post-SOT), Visit 13 (3-months post-SOT), Visit 14 (6-months post-SOT), and Visit 16 (12-months post-SOT)
Population: Per Protocol Set presented. Data were not available for one Group 1 subject at Visit 14, three Group 1 subjects at Visit 16, and one Group 2 subject at Visit 7. In accordance with the planned study protocol, Group 2 subjects were not assessed for this outcome at 6- and 12-months due to crossover to receive active stimulation.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 13 | 16
Participants
  Visit 7: 4-weeks Post-SOT: number analyzed (Participants) | 13 | 15
  Visit 7: 4-weeks Post-SOT | 7 | 6
  Visit 11: 8-weeks Post-SOT | 10 | 8
  Visit 13: 3-months Post-SOT | 10 | 6
  Visit 14: 6-months Post-SOT: number analyzed (Participants) | 12 | 0
  Visit 14: 6-months Post-SOT | 9 |
  Visit 16: 12-months Post-SOT: number analyzed (Participants) | 10 | 0
  Visit 16: 12-months Post-SOT | 6 |

4. Secondary Outcome: Pain Disability Index (PDI)
Description: The Pain Disability Index (PDI) is a validated survey measuring the degree to which pain disrupts 7 categories of life activities on a scale from 0 to 10, with higher scores indicating greater disability. The 7 scores were summed for each subject to provide an overall pain disability score ranging from 0 to 70. A score of 0 indicates no disability while a score of 70 signifies that all of the activities in which the individual would normally be involved have been totally disrupted or prevented by pain. To be considered a success, subjects must have a ≥ 10-point reduction in their total PDI score at each time point compared to their baseline score. The number of subjects successful at each time point is reported.
Time Frame: as for outcome 3
Population: Per Protocol Set presented. Data were not available for one Group 2 subject at Visit 7, one Group 1 subject at Visit 14, and three Group 1 subjects at Visit 16. In accordance with the planned study protocol, Group 2 subjects were not assessed for this outcome at 6- and 12-months due to crossover to receive active stimulation.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 13 | 16
Participants
  Visit 7: 4-weeks Post-SOT: number analyzed (Participants) | 13 | 15
  Visit 7: 4-weeks Post-SOT | 10 | 9
  Visit 11: 8-weeks Post-SOT | 10 | 9
  Visit 13: 3-months Post-SOT | 12 | 5
  Visit 14: 6-months Post-SOT: number analyzed (Participants) | 12 | 0
  Visit 14: 6-months Post-SOT | 10 |
  Visit 16: 12-months Post-SOT: number analyzed (Participants) | 10 | 0
  Visit 16: 12-months Post-SOT | 6 |

5. Secondary Outcome: Patient Global Impression of Change (PGIC) Survey
Description: The Patient Global Impression of Change (PGIC) Survey asks subjects to rate their improvement with treatment on a 7-point scale ranging from -3 to 0 to +3, where -3 represents "very much worse," 0 is "no change," and +3 represents "very much improved" as compared to before stimulation treatment. The subjects combine all the components of their experience into one overall score. The mean rank score of each group was calculated for each time frame.
Time Frame: Visit 7 (4-weeks post-Start of Therapy [SOT]), Visit 11 (8-weeks post-SOT), Visit 13 (3-months post-SOT), Visit 14 (6-months post-SOT), and Visit 16 (12-months post-SOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 13 | 16
score on a scale
  Visit 7: 4-weeks Post-SOT: number analyzed (Participants) | 13 | 15
  Visit 7: 4-weeks Post-SOT | 1.8 (0.73) | 1.0 (1.1)
  Visit 11: 8-weeks Post-SOT | 1.5 (0.66) | 0.88 (1.6)
  Visit 13: 3-months Post-SOT | 1.2 (0.93) | 0.75 (1.2)
  Visit 14: 6-months Post-SOT: number analyzed (Participants) | 12 | 0
  Visit 14: 6-months Post-SOT | 1.3 (1.4) |
  Visit 16: 12-months Post-SOT: number analyzed (Participants) | 10 | 0
  Visit 16: 12-months Post-SOT | 1.3 (1.3) |

6. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: The Pain Catastrophizing Scale (PCS) questionnaire has 13 questions that assess rumination, magnification, and helplessness. Subjects are asked to think back on painful experiences in the past and reflect on how often they had specific thoughts or feelings. Each of the 13 questions is scored on a 5-point scale where 0 represents "not at all," and 4 represents "all the time." The scores from each question were summed for each subject to provide a total PCS score, with a possible range from 0 to 52 with higher scores indicating a greater tendency to catastrophize pain (i.e. a higher score indicates a worse outcome). The mean score for each time point is presented.
Time Frame: Visit 1 (Baseline), Visit 7 (4-weeks post-Start of Treatment [SOT]), and Visit 11 (8-weeks post-SOT)
Population: Per Protocol Set presented. Data were not available for one Group 2 subject at Visit 7.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 13 | 16
score on a scale
  Visit 1: Baseline | 17.6 (10.1) | 24.1 (11.6)
  Visit 7: 4-weeks Post-SOT: number analyzed (Participants) | 13 | 15
  Visit 7: 4-weeks Post-SOT | 12.3 (10.0) | 17.2 (14.3)
  Visit 11: 8-weeks Post-SOT | 8.3 (8.4) | 19.2 (15.4)

7. Secondary Outcome: Pain Medication Usage
Description: Subjects completed 7-day diaries in which they tracked their daily use of analgesic medications. Opioid analgesic usage was converted into a morphine equivalent dosage (MED), which is measured in units of morphine milligram equivalents (MME), for subjects who were using opioid analgesics at baseline. The average MED was calculated for each subject at each time point.
Time Frame: Baseline, 1 to 4 weeks post-start of treatment (SOT), 5 to 8 weeks post-SOT, 3 months post-SOT, 6 months post-SOT, and 12 months post-SOT
Population: Per protocol set presented; only the six subjects that were using opioid analgesics at baseline were included in the analysis. Data were not available for two Group 1 subjects at 12-months post-SOT and for one Group 2 subject at 3-months post-SOT. In accordance with the planned study protocol, Group 2 subjects were not assessed for this outcome at 6- and 12-months due to crossover to receive active stimulation.
Measure: Mean (Standard Deviation); unit: MME (Morphine Milligram Equivalents)
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 3 | 3
MME (Morphine Milligram Equivalents)
  Baseline | 32.3 (37.2) | 14.4 (13.7)
  1 to 4 weeks Post-SOT | 32.4 (36.9) | 16.3 (13.0)
  5 to 8 weeks Post-SOT | 30.4 (38.7) | 12.4 (10.4)
  3-months Post-SOT: number analyzed (Participants) | 3 | 2
  3-months Post-SOT | 30.7 (38.9) | 9.0 (12.7)
  6-months Post-SOT: number analyzed (Participants) | 3 | 0
  6-months Post-SOT | 21.1 (21.5) |
  12-months Post-SOT: number analyzed (Participants) | 1 | 0
  12-months Post-SOT | 45.0 (0.0) |

8. Secondary Outcome: Number of Subjects With ≥ 50% Reduction in Average Post-Amputation Pain (Residual Limb Pain [RLP] and/or Phantom Limb Pain [PLP]) 1 to 4 Weeks After Start of Treatment
Description: All subjects were asked to complete daily diaries to record their average residual limb pain and/or phantom pain intensities during the past 24 hours on each day of a 7-day period using an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average pain scores were calculated across the 7-day period for each region of pain at baseline and across weeks 1 to 4 post-start of treatment (i.e., the first half of the 8-week treatment period). Percent reduction was then calculated for each subject's qualifying region of pain (residual limb and/or phantom limb pain with qualifying average pain intensity at baseline). To be considered a success, subjects must have experienced ≥ 50% reduction in all qualifying regions of pain compared to their 7-day baseline diary average pain score(s). The number of successes is presented.
Time Frame: Baseline and 1 to 4 weeks post-start of treatment (SOT)
Population: Per Protocol Set presented. One Group 2 subject only had 3 days of diary data during week 3 post-SOT.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 13 | 16
Participants | 3 | 3

9. Secondary Outcome: Number of Subjects With ≥ 50% Reduction in Average Residual Limb Pain (RLP) 5 to 8 Weeks After Start of Treatment
Description: All subjects were asked to complete daily diaries to record their average residual limb pain and/or phantom pain intensities during the past 24 hours on each day of a 7-day period using an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average residual limb pain scores were calculated across the 7-day period at baseline and for weeks 5 to 8 post-start of treatment (for subjects with qualifying residual limb average pain intensity at baseline). Percent reduction from baseline was then calculated, and the number of subjects that experienced ≥ 50% reduction in residual limb pain are reported.
Time Frame: Baseline and 5 to 8 weeks post-start of treatment (SOT)
Population: Per Protocol Set of subjects that qualified with residual limb pain presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 10 | 13
Participants | 5 | 3

10. Secondary Outcome: Number of Subjects With ≥ 50% Reduction in Average Phantom Limb Pain (PLP) 5 to 8 Weeks After Start of Treatment
Description: All subjects were asked to complete daily diaries to record their average residual limb pain and/or phantom pain intensities during the past 24 hours on each day of a 7-day period using an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average phantom limb pain scores were calculated across the 7-day period at baseline and for weeks 5 to 8 post-start of treatment (for subjects with qualifying phantom limb average pain intensity at baseline). Percent reduction from baseline was then calculated, and the number of subjects that experienced ≥ 50% reduction in phantom limb pain are reported.
Time Frame: Baseline and 5 to 8 weeks post-start of treatment (SOT)
Population: Per Protocol Set of subjects that qualified with phantom limb pain presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 12 | 14
Participants | 7 | 3

11. Secondary Outcome: Durability of Treatment Effect on Average Post-Amputation Pain Intensity (Residual Limb Pain [RLP] and/or Phantom Limb Pain [PLP])
Description: All subjects were asked to complete daily diaries to record their average residual limb pain and/or phantom limb pain intensities during the past 24 hours on each day of a 7-day period using an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average pain scores were calculated across the 7-day period for each region of pain at baseline and at 3, 6, and 12 months post-start of treatment. Percent reduction was then calculated for each subject's qualifying region of pain (residual limb and/or phantom limb pain with qualifying average pain intensity at baseline) at each time point. To be considered a success, subjects must have experienced ≥ 50% reduction in all qualifying regions of pain compared to their 7-day baseline diary average pain score(s). The number of successes is presented.
Time Frame: Baseline, 3-months post-Start of Treatment (SOT), 6-months post-SOT, and 12-months post-SOT
Population: Per Protocol Set presented. Data were not available for one Group 1 subject at 6-months and for three at 12-months. In accordance with the planned study protocol, Group 2 subjects were not assessed for this outcome at 6- and 12-months due to crossover to receive active stimulation.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 13 | 16
Participants
  3-months Post-SOT | 4 | 3
  6-months Post-SOT: number analyzed (Participants) | 12 | 0
  6-months Post-SOT | 4 | 0
  12-months Post-SOT: number analyzed (Participants) | 10 | 0
  12-months Post-SOT | 3 | 0

ADVERSE EVENTS:
Time Frame: Each participant enrolled was assessed for adverse events from the time of informed consent through their final study visit. For subjects in Group 1, the total assessment period was approximately 14 months for each participant. Each Group 2 subject that did not crossover to receive stimulation treatment was assessed for approximately 5 months. Group 2 subjects that crossed over to receive treatment were each assessed for approximately 18 months.
Groups:
- Group 2 (Control Group Treatment Crossover): Subjects who were consented and randomized to Group 2 (Control), received sham stimulation treatment, and crossed over to receive active stimulation treatment.
Arm/Group | Group 1 (Treatment) | Group 2 (Control) | Group 2 (Control Group Treatment Crossover)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/9
Other Adverse Events (participants affected / at risk) | 10/19 | 6/19 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Treatment) (N=19) | Group 2 (Control) (N=19) | Group 2 (Control Group Treatment Crossover) (N=9)
Skin irritation (Skin and subcutaneous tissue disorders) | 7 (9) | 5 (6) | 2 (2)
Itching at bandage site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Discoloration/bruising (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin tear at pad site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain at lead site (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Uncomfortable stimulation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT03783689/Prot_002.pdf
  • Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03783689/SAP_003.pdf